CLINICAL TRIAL: NCT06735521
Title: Att Överleva Och Leva Som Vuxen Med Enkammarhjärta I Sverige
Brief Title: Cardiac Magnetic Resonance Stress-perfusion Study in Patinets with Fontan Circulation
Acronym: CMR_TCPC
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Peder Sörensson, Senior Consultant in Cardiology, Karolinska Institutet
Other Study IDs: Dnr 2022-04574-01
Record Dates: First submitted 2024-10-16; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Univentricular Heart; Microvascular Dysfunction; Heart Failure; Magnetic Resonance
Keywords: Fontan circulation; CMR; stress-perfusion; tissue characterization; univentricle heart; TCPC
MeSH Terms: conditions — Univentricular Heart; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Univentricle heart, operated with TCPC (total cavo pulmonary connection)
  Interventions: Diagnostic Test: Cardiac magnetic resonance stress-perfusion

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance stress-perfusion — Included patients will be examined at the Karolinska University Hospital in a 1.5T Siemens Sola magnetic resonance camera at rest and during adenosine stress with specific CMR sequences (adenosine stress-perfusion, myocardial velocities, and tissue characterization) for non-invasive determination of macro- and microvascular dysfunction, global myocardial function, pulmonary artery pressure and scarring of the myocardium.
  Adenosine or Regadenoson will be used as stress medication which is according to clinical routine. Adenosine will be infused over approximately 5 minutes (110-140 μg / kg/min), Regadenoson (5 ml) will be a 10-second injection (400 μg single dosage). Intravenous gadolinium-based contrast agents will be administered, Gadovist (1 mmol/ml, gadobuterol), 0.15 mmol/kg during stress and rest.

SUMMARY:
Univentricular heart (UVH) is a severe congenital heart disease. Accurate advanced non-invasive diagnostic methods is limited. Cardiovascular magnetic resonance (CMR) imaging has evolved as a particularly useful tool for the study of patients with adult congenital heart disease (ACHD) considering its ability to determine detailed anatomy and detect early cardiac dysfunction without the need for radiation exposure. Most of contemporary treatment recommendations are based on consensus opinions/documents and small studies from local, or national registries. Improved knowledge is needed in all these areas to facilitate clinical decisions regarding treatment, monitoring and follow-up.

This study seeks to answer if early detection of deterioration in cardiac function, venous pressure and microvascular dysfunction can identify patients before the symptoms progress and thus help to initiate early treatment. The hypothesis is that quantitative myocardial stress-perfusion maps improves the pathophysiological insight in patients with UVH.

The overall goal with this research proposal is to implement combined advanced CMR imaging for a comprehensive non-invasive mapping of functional cardiovascular behavior in patients with complex UVH disease. The outcome of this research may benefit this young adult patient population due to early detection of cardiac disease, less hospitalizations because of heart failure, and eventually decrease morbidity and mortality.

DETAILED DESCRIPTION:
CMR is performed supine with a Magnetom Aera® 1.5 Tesla (T) scanner (Siemens Healthcare, Erlangen, Germany), with a phased-array 18-channel body matrix coil and a spine matrix coil. A venous blood sample is drawn to determine hematocrit and blood creatinine prior to imaging. Full coverage retrospective electrocardiographic (ECG)-gated balanced steady state free precession (bSSFP) cine imaging is acquired in standard three long-axis and short-axis slices. Typical imaging parameters are flip angle 68°, pixel size 1.4 × 1.9 mm2, slice thickness 8.0 mm, echo time (TE)/repetition time (TR) 1.19/37.05 ms, matrix size 256 × 144 and field of view (FOV) 360 × 270 mm2.

Using first-pass perfusion imaging, quantitative perfusion maps (ml/min/g) are acquired in one short-axis and one long-axis slice (mid-ventricular, 2-chamber) during administration of an intravenous contrast-agent bolus (0.05 mmol/kg, gadobutrol, Gadovist, Bayer AB, Solna, Sweden), during adenosine infusion (110 µg/kg/min or increased according to clinical routine to 140 µg/kg/min in the absence of adequate response to adenosine (Adenosine, Life Medical AB, Stockholm) and in subsequent rest. Adenosine response is assessed clinically based on symptoms and heart rate response. Adenosine and contrast agent are administered in two different cannulas. Subjects abstained from caffeine for 24 hours prior to CMR examination. A distributed tissue exchange model is used to compute the perfusion maps and the Gadgetron (reconstruction computer) inline perfusion mapping software is used to generate the perfusion maps.Typical imaging parameters were bSSFP single shot readout, flip angel 50°, slice thickness 8.0 mm, TE/TR 1.04/2.5 ms, bandwidth 1085 Hz/pixel, FOV 360 × 270 mm2 and saturation delay/trigger delay (TD) 95/40 ms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had undergone total cavo-pulmonary connection (TCPC) surgery resulting in Fontan circulation.
* NYHA (New York Heart Assosiation) class I-II.
* Understanding the study information (signed informed consent).
* >18 years old.

Exclusion Criteria:

* Device therapy (pacemaker, ICD).
* Failing Fontan (NYHA III-IV).
* Kidney failure (GFR<30ml/h).
* Arrythmia (atrial fibrillation).
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The project is planned as a prospective cohort study where approximately 30 patients with Fontan circulation will be included. The cohort is out-clinic patients at the tertiary adult congenital heart disease center at the Karolinska University Hospital in Stockholm, Sweden. The patients will be asked to participate in the study when they have a clinical visit at Karolinska by the treating physician or nurse. Inclusion and exclusion criteria are shown above.
  Additional data will be collected from the patient cohort; age, gender, underlying diagnoses, interventions, medication, symptoms, NYHA functional class, ECG, cardiac pulmonary exercise results, self-reported level of physical activity, pacemaker / implantable cardioverter defibrillator (ICD), and quality of life assessed by EuroQoL 5-dimensional questionnaire (EQ-5D).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Detection of microvascular dysfunction in patients with UVH | Through study completion, an average of 1 year
  This project aims to evaluate microvascular dysfunction using quantitative stress-perfusion CMR in patients with different morphological systemic chamber (left vs right).

SECONDARY OUTCOMES:
To detect and compare tissue characterization. | Through study completion, an average of 1 year
  Investigate whether positive findings in tissue characterization is higher in different systemic ventricles (left vs right) using T1 and T2-mapping, LGE (late gadolinium enhancement, myocardial scar).

OTHER OUTCOMES:
Venous pressure in TCPC | Through study completion, an average of 1 year
  Calculate venous delta pressure (customized in-house software) in the cavo-pulmonary connection using CMR 4D-flow imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
IPD used i the results publication.
Supporting Information: Study Protocol, CSR
Time Frame: April 2024 - April 2026.
Access Criteria: On written request to the PI from researchers in the same field of interests.

REFERENCES:
- [Background] Rychik J, Atz AM, Celermajer DS, Deal BJ, Gatzoulis MA, Gewillig MH, Hsia TY, Hsu DT, Kovacs AH, McCrindle BW, Newburger JW, Pike NA, Rodefeld M, Rosenthal DN, Schumacher KR, Marino BS, Stout K, Veldtman G, Younoszai AK, d'Udekem Y; American Heart Association Council on Cardiovascular Disease in the Young and Council on Cardiovascular and Stroke Nursing. Evaluation and Management of the Child and Adult With Fontan Circulation: A Scientific Statement From the American Heart Association. Circulation. 2019 Aug 6;140(6):e234-e284. doi: 10.1161/CIR.0000000000000696. Epub 2019 Jul 1. PMID 31256636
- [Background] Di Salvo G, Miller O, Babu Narayan S, Li W, Budts W, Valsangiacomo Buechel ER, Frigiola A, van den Bosch AE, Bonello B, Mertens L, Hussain T, Parish V, Habib G, Edvardsen T, Geva T, Baumgartner H, Gatzoulis MA; 2016-2018 EACVI Scientific Documents Committee. Imaging the adult with congenital heart disease: a multimodality imaging approach-position paper from the EACVI. Eur Heart J Cardiovasc Imaging. 2018 Oct 1;19(10):1077-1098. doi: 10.1093/ehjci/jey102. PMID 30084968
- [Background] Dalen M, Odermarsky M, Liuba P, Johansson Ramgren J, Synnergren M, Sunnegardh J. Long-Term Survival After Single-Ventricle Palliation: A Swedish Nationwide Cohort Study. J Am Heart Assoc. 2024 Mar 19;13(6):e031722. doi: 10.1161/JAHA.123.031722. Epub 2024 Mar 18. PMID 38497454